CLINICAL TRIAL: NCT02766322
Title: Pharmacokinetics and Subjective Responses to Alcohol After Bariatric Surgery
Brief Title: Alcohol and Bariatric Surgery
Acronym: ABS
Status: Terminated | Type: Observational
Why Stopped: Recruitment affected by COVID, then grant ended
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Carle Foundation Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 16135; 17205 (Other: UIUC)
Record Dates: First submitted 2016-04-27; First posted 2016-05-09 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Alcohol metabolism; Bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Ethanol; Constriction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and Plasma
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (7):
- Gastric Bypass longitudinal: Morbidly obese subjects undergoing gastric bypass surgery. Subjects will be assessed in four testing sessions about 1 week apart in a randomized cross-over fashion before surgery. During the first two sessions, their response to alcohol or nonalcoholic (placebo) beverage will be evaluated. During testing sessions three and four, their response to alcohol administered intravenously will be evaluated. These four testing sessions will be repeated when subjects loose ~ 16% of their presurgery body weight.
  Interventions: Other: Oral Alcohol challenge test Alcohol visit first; Other: Oral Alcohol challenge test Placebo visit first; Other: Intravenous Alcohol Challenge Test (Clamp); Other: Intravenous Alcohol Self-administration Test
- Gastric Banding longitudinal: Morbidly obese subjects undergoing laparoscopic gastric banding surgery. Subjects will be assessed in four testing sessions about 1 week apart in a randomized cross-over fashion before surgery. During the first two sessions, their response to alcohol or nonalcoholic (placebo) beverage will be evaluated. During testing sessions three and four, their response to alcohol administered intravenously will be evaluated. These four testing sessions will be repeated when subjects loose ~ 16% of their presurgery body weight.
  Interventions: Other: Oral Alcohol challenge test Alcohol visit first; Other: Oral Alcohol challenge test Placebo visit first; Other: Intravenous Alcohol Challenge Test (Clamp); Other: Intravenous Alcohol Self-administration Test
- Sleeve gastrectomy longitudinal: Morbidly obese subjects undergoing sleeve gastrectomy surgery. Subjects will be assessed in four testing sessions about 1 week apart in a randomized cross-over fashion before surgery. During the first two sessions, their response to alcohol or nonalcoholic (placebo) beverage will be evaluated. During testing sessions three and four, their response to alcohol administered intravenously will be evaluated. These four testing sessions will be repeated when subjects loose ~ 16% of their presurgery body weight..
  Interventions: Other: Oral Alcohol challenge test Alcohol visit first; Other: Oral Alcohol challenge test Placebo visit first; Other: Intravenous Alcohol Challenge Test (Clamp); Other: Intravenous Alcohol Self-administration Test
- Gastric Bypass (cross-sectional): Subjects who underwent gastric bypass surgery 1-5 years ago. Subjects will be assessed in four testing sessions about 1 week apart in a randomized cross-over fashion after surgery. During the first two sessions, their response to alcohol or nonalcoholic (placebo) beverage will be evaluated. During testing sessions three and four, their response to alcohol administered intravenously will be evaluated.
  Interventions: Other: Oral Alcohol challenge test Alcohol visit first; Other: Oral Alcohol challenge test Placebo visit first; Other: Intravenous Alcohol Challenge Test (Clamp); Other: Intravenous Alcohol Self-administration Test
- Gastric Banding (cross-sectional): Subjects who underwent gastric banding surgery 1-5 years ago. Subjects will be assessed in four testing sessions about 1 week apart in a randomized cross-over fashion after surgery. During the first two sessions, their response to alcohol or nonalcoholic (placebo) beverage will be evaluated. During testing sessions three and four, their response to alcohol administered intravenously will be evaluated.
  Interventions: Other: Oral Alcohol challenge test Alcohol visit first; Other: Oral Alcohol challenge test Placebo visit first; Other: Intravenous Alcohol Challenge Test (Clamp); Other: Intravenous Alcohol Self-administration Test
- Sleeve gastrectomy (cross-sectional): Subjects who underwent sleeve gastrectomy surgery 1-5 years ago. Subjects will be assessed in four testing sessions about 1 week apart in a randomized cross-over fashion after surgery. During the first two sessions, their response to alcohol or nonalcoholic (placebo) beverage will be evaluated. During testing sessions three and four, their response to alcohol administered intravenously will be evaluated.
  Interventions: Other: Oral Alcohol challenge test Alcohol visit first; Other: Oral Alcohol challenge test Placebo visit first; Other: Intravenous Alcohol Challenge Test (Clamp); Other: Intravenous Alcohol Self-administration Test
- Non-surgical group: Subjects who are age and body mass index equivalent to gastric bypass (cross-sectional) and Sleeve gastrectomy (cross-sectional) but did not undergo any type of bariatric surgery. Subjects will be assessed in four testing sessions about 1 week apart in a randomized cross-over fashion after surgery. During the first two sessions, their response to alcohol or nonalcoholic (placebo) beverage will be evaluated. During testing sessions three and four, their response to alcohol administered intravenously will be evaluated.
  Interventions: Other: Oral Alcohol challenge test Alcohol visit first; Other: Oral Alcohol challenge test Placebo visit first; Other: Intravenous Alcohol Challenge Test (Clamp); Other: Intravenous Alcohol Self-administration Test

INTERVENTIONS:
Other: Oral Alcohol challenge test Alcohol visit first — Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion (visit 1 alcohol, visit 2 placebo).
Other: Oral Alcohol challenge test Placebo visit first — Subjects will be assessed in two testing sessions about 1 week apart, in which their response to alcohol or nonalcoholic (placebo) beverage will be evaluated in a randomized cross-over fashion (visit 1 placebo, visit 2 alcohol).
Other: Intravenous Alcohol Challenge Test (Clamp) — Subjects will be evaluated with an alcohol clamp (i.e. alcohol will be infused intravenously until reaching 60mg/dl and this blood alcohol concentration will be kept constant for two hours). We will record subjective responses to alcohol throughout different times of the clamp.
Other: Intravenous Alcohol Self-administration Test — Subjects will be asked to press a button ("work") to receive either a "drink" or saline through an IV catheter. The amount of alcohol infused after earning their reward will be based on their body composition and will raise their blood alcohol level by 10 mg/dl (eight time less than the legal limit for driving). We will set a safety limit to 150 mg/dl so that subjects will not be allowed to work for alcohol until their blood alcohol levels go below that limit.

SUMMARY:
The investigators wish to study the effects of alcohol on three forms of bariatric surgery, Roux-en-Y gastric bypass (RYGB), sleeve gastrectomy (SG) and laparoscopic adjustable gastric banding (LAGB) and compare them with a non-surgical group. The surgery is not part of the clinical trial. If insurance does not cover the procedure, then the patient is responsible for payment of the surgical process. The investigators are doing pre and post surgery testing to provide a better understanding of the effect of bariatric surgery-induced weight loss on 1) alcohol absorption, distribution and elimination from the body, 2) the effects of alcohol on mood, and 3) the effects of alcohol on driving.

DETAILED DESCRIPTION:
The study includes seven groups of women: One group will be undergoing RYGB another group will be undergoing LAGB, a third group will be undergoing SG, the fourth group will be women who underwent RYGB 1-5 years ago, the fifth group will be women who underwent LAGB 1-5 years ago, the sixth group will be women who underwent SG 1-5 years ago and the seventh group will be women who have equivalent age and body mass index than women in the groups who underwent RYGB or SG 1-5 years ago but did not have bariatric surgery (non-surgical group).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Drink at least 1 standard alcoholic beverage/ month
* Underwent RYGB, SG, or LAGB 1-5 years ago or will undergo RYGB, SG, or LAGB surgery
* Did not undergo bariatric surgery (for the non-surgical group)

Exclusion Criteria:

* Male
* Smoker or quit < 6 months ago
* Anemia
* Liver disease
* Body weight > 450 pounds
* Taking medications that can interact with alcohol metabolism or the subjective effects of alcohol

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Bariatric surgery clinic
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Change in the peak blood alcohol level achieved before-after bariatric surgery and among bariatric surgery and control groups | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  Time to reach peak blood alcohol levels and height of blood alcohol levels will be examined before and after surgery and compared between those who had gastric bypass or gastric sleeve versus lap banding and the non-surgery control group.
Change in alcohol subjective effects from pre- to post- bariatric surgery and among bariatric surgery and control groups | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  Validated instruments (such as the Addiction Research Center Inventory and the biphasic alcohol effect scale) will be used to measure alcohol's subjective effects at different timepoints after drinking an alcoholic or a non-alcoholic (control) beverage as well as receiving alcohol vs placebo orally or alcohol intravenously
Change in the area under the curve for blood alcohol concentration (BAC) versus time pre- to post-bariatric surgery and among different bariatric surgery groups and controls | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  The area under the curve for BAC will be examined before and after surgery and compared among those who had gastric bypass or gastric sleeve versus lap banding or the non-surgery control group.
Change in the rate of alcohol elimination between pre- and post-surgery and among the different bariatric surgery groups and the control groups. | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  The systemic alcohol elimination rate calculated from the alcohol infusion rate during the iv alcohol clamp technique will be compared pre- to post- surgery and among bariatric and control groups

SECONDARY OUTCOMES:
Changes in alcohol's effects on glucose homeostasis [pre- to post-surgery and among bariatric surgery groups and control groups. | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  mmol/L
Changes in alcohol's effects on insulin [pre- to post-surgery and among bariatric surgery groups and control groups. | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  pmol/L
Changes in alcohol's effects on C-peptide [pre- to post-surgery and among bariatric surgery groups and control groups. | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  nmol/L
Changes in alcohol's effects on FGF21 [pre- to post-surgery and among bariatric surgery groups and control groups. | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  pg/ml
Changes in alcohol's effects on ghrelin [pre- to post-surgery and among bariatric surgery groups and control groups. | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  pg/ml
Changes in alcohol's effects on GLP-1 [pre- to post-surgery and among bariatric surgery groups and control groups. | Subjects in the longitudinal arm of the study will be assessed before surgery and approximately 9 months after surgery. A group of subjects will be assessed 1-5 years after surgery only.
  pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Marta Y Pepino de Gruev, PhD, Principal Investigator — UIUC
Locations (1):
- University of Illinois at Urbana Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Seyedsadjadi N, Acevedo MB, Alfaro R, Ramchandani VA, Plawecki MH, Rowitz B, Pepino MY. Site of Alcohol First-Pass Metabolism Among Women. JAMA Netw Open. 2022 Mar 1;5(3):e223711. doi: 10.1001/jamanetworkopen.2022.3711. PMID 35315921
- [Background] Acevedo MB, Teran-Garcia M, Bucholz KK, Eagon JC, Bartholow BD, Burd NA, Khan N, Rowitz B, Pepino MY. Alcohol sensitivity in women after undergoing bariatric surgery: a cross-sectional study. Surg Obes Relat Dis. 2020 Apr;16(4):536-544. doi: 10.1016/j.soard.2020.01.014. Epub 2020 Jan 23. PMID 32075778
- [Background] Acevedo MB, Eagon JC, Bartholow BD, Klein S, Bucholz KK, Pepino MY. Sleeve gastrectomy surgery: when 2 alcoholic drinks are converted to 4. Surg Obes Relat Dis. 2018 Mar;14(3):277-283. doi: 10.1016/j.soard.2017.11.010. Epub 2017 Nov 10. PMID 29305304
- [Background] Seyedsadjadi N, Ramchandani VA, Plawecki MH, Kosobud AEK, O'Connor S, Rowitz B, Pepino MY. Fat-free mass accounts for most of the variance in alcohol elimination rate in women. Alcohol Clin Exp Res (Hoboken). 2023 May;47(5):848-855. doi: 10.1111/acer.15047. Epub 2023 Mar 14. PMID 36871954
- [Background] Seyedsadjadi N, Ramchandani VA, Plawecki MH, Kosobud AEK, O'Connor S, Rowitz B, Pepino MY. Response to commentary on: "Fat-free mass accounts for most of the variance in alcohol elimination rate in women". Alcohol Clin Exp Res (Hoboken). 2023 Sep;47(9):1646-1648. doi: 10.1111/acer.15142. Epub 2023 Jul 11. No abstract available. PMID 37407434
- [Derived] Molina-Castro M, Rowitz B, Pepino MY. Glucagon-like peptide-1, fibroblast growth factor 21, and other endocrine responses to alcohol ingestion in women before and after metabolic surgery. Front Pharmacol. 2025 May 22;16:1575156. doi: 10.3389/fphar.2025.1575156. eCollection 2025. PMID 40474966